CLINICAL TRIAL: NCT00178490
Title: Neurocognitive Function in Children With Hypertension
Brief Title: Effect of High Blood Pressure and Antihypertensive Treatment on Brain Functioning in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marc Lande, Professor, University of Rochester
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 550; K23HL080068 (NIH); 10361
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
Keywords: Neurocognitive Function
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Children with high blood pressure who will receive treatment for high blood pressure
  Interventions: Drug: High blood pressure treatment
- 2 (No Intervention): Children with normal blood pressure who will undergo no treatment

INTERVENTIONS:
Drug: High blood pressure treatment — Participants who are identified as having high blood pressure will be given by a pediatric nephrologist a 12-month treatment plan for their high blood pressure. The treatment plan will include a combination of diet, weight loss, increased exercise, and if needed, blood pressure medication. Participants receiving medication treatment will be treated with a calcium channel blocker and/or ACE inhibitor.
  Arms: 1

SUMMARY:
High blood pressure, or hypertension, affects up to 10% of minority children and adolescents. Although complications of high blood pressure, such as stroke and heart attack, are uncommon in childhood, high blood pressure-related organ damage can occur at a young age. Studies with young adults have indicated that high blood pressure can affect the central nervous system, resulting in deficits in brain function. However, more research is necessary to confirm the association between neurocognitive deficits and high blood pressure in children and to determine if these deficits are reversible with treatment. This study will determine whether high blood pressure in children and adolescents has subtle effects on learning, attention, and concentration. The study will also determine the effect of an antihypertensive treatment plan, involving a combination of diet, weight loss, increased exercise, and if needed, blood pressure medication, on brain function in children and adolescents receiving treatment for high blood pressure.

DETAILED DESCRIPTION:
High blood pressure is a condition that normally affects adults, but can affect young children and adolescents, as well. High blood pressure in children is most commonly caused by unhealthy lifestyle or family history, but it can also be due to disease, such as kidney or heart disease. When a person has high blood pressure, the heart must work harder to pump blood throughout the body. If left untreated, high blood pressure can eventually cause damage to the heart, kidneys, and eyes. Recent studies have linked high blood pressure in children to deficits in brain functioning. However, more information is needed to confirm this connection and to determine the effectiveness of antihypertensive treatments in restoring brain function. This study will determine the effect of high blood pressure on brain functioning in children and adolescents. The study will also determine the effect of an antihypertensive treatment plan, involving a combination of diet, weight loss, increased exercise, and if needed, blood pressure medication, on brain function in children and adolescents receiving treatment for high blood pressure.

Participation in this study will last 12 months and will involve children with high blood pressure and children with normal blood pressure. Information on participants' medical history and sleep patterns, as well as parent's income and education level, will be collected. Participants with suspected high blood pressure will then undergo 24-hour blood pressure monitoring using an ambulatory blood pressure cuff. Afterwards, participants who are determined to have high blood pressure will undergo an echocardiogram of the heart. These participants will soon return to the General Clinical Research Center (GCRC) to undergo additional testing, which will include measurements of height, weight, and body mass index; a urine sampling; and a blood draw.

Before beginning potential treatment, both healthy and high blood pressure participants will complete a series of thinking and learning tests that will take about 90 minutes. Parents of participants will also be asked to answer a 10-minute questionnaire about their child's behavior and emotions. Participants with high blood pressure will then start a 12-month antihypertensive treatment plan, which will involve a combination of diet, weight loss, increased exercise, and if needed, blood pressure medication. A digital blood pressure cuff will be provided to participants for at-home blood pressure monitoring. During the treatment period, a study nurse will call participants every 1 to 2 weeks for the first 3 months and monthly for the remaining 9 months to check on blood pressure readings and to refill medications. Participants will be seen at the GCRC once every 3 to 4 months to monitor and adjust treatment as needed. Healthy participants will undergo no study treatment during the treatment phase.

Upon completion of the 12 months of treatment, all participants will undergo repeat thinking and learning tests, and parents of participants will complete repeat questionnaires. Participants with high blood pressure will also repeat the 24-hour blood pressure monitoring test.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* No known learning disorder, disorders of cognitive function, treatment with medications for attention deficit, or history of severe head injury (loss of consciousness for more than 30 minutes)
* Casual blood pressure greater than or equal to 90th percentile for age, gender, and height during clinic visit and on at least two other previous occasions

Exclusion Criteria:

* Secondary cause of high blood pressure
* Chronic disease
* History of treatment for elevated lead level
* History of maternal substance use during pregnancy
* Evidence of obstructive sleep apnea

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Neurocognitive function improvement with normalization of blood pressure | Measured at Month 12

SECONDARY OUTCOMES:
Treatment of hypertension | Measured at Month 12
Correlation of neurocognitive deficits with the presence of cardiac hypertrophy, microalbuminuria, and hypertensive retinopathy | Measured at Month 12
Correlation of the presence of neurocognitive deficits with severity and pattern of hypertension | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Marc B. Lande, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Strong Memorial Hospital, Rochester, New York, United States

REFERENCES:
- [Background] Lande MB, Kaczorowski JM, Auinger P, Schwartz GJ, Weitzman M. Elevated blood pressure and decreased cognitive function among school-age children and adolescents in the United States. J Pediatr. 2003 Dec;143(6):720-4. doi: 10.1067/S0022-3476(03)00412-8. PMID 14657815
- [Background] Miller RE, Shapiro AP, King HE, Ginchereau EH, Hosutt JA. Effect of antihypertensive treatment on the behavioral consequences of elevated blood pressure. Hypertension. 1984 Mar-Apr;6(2 Pt 1):202-8. PMID 6724662